CLINICAL TRIAL: NCT05748769
Title: Ipsilateral Transfer of Motor Skill From Upper to Lower Limb in Healthy Adults: a Randomized Controlled Trial
Brief Title: Ipsilateral Transfer of Motor Skill From Upper to Lower Limb in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AU-HEA-OE-20210610-B
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: ipsilateral transfer; motor performance; Upper limb; Lower limb; reaching sequence
MeSH Terms: interventions — Observation

STUDY DESIGN:
Intervention Model Description: Randomized control trial (RCT)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UL group (Experimental): SIngle session of practicing RM sequence with the UL towards illuminating switches
  Interventions: Behavioral: Practice (UL)
- Switches observation - SO group (Active Comparator): Single session of observation of sequence of illuminating switches
  Interventions: Behavioral: Observation (SO)
- (Nature observation -NO group (Active Comparator): Single session of observation of nature movies
  Interventions: Behavioral: Nature Observation (NO)

INTERVENTIONS:
Behavioral: Practice (UL) — Subjects performed RMs toward the units that were activated in the same order as the tested sequence 1-4-3-5-4-2, and with an activation duration and delay of 1 s. The practice included 16 blocks, each consisting of 30 RM with a 30 s pause after each block
  Arms: UL group
Behavioral: Observation (SO) — Subjects observed the illuminating switches while avoiding moving. The subjects observed RMs toward the units that were activated in the same order as the practiced sequence 1-4-3-5-4-2, also with an activation duration and delay of 1 s and 30 s pause after each block.
  Arms: Switches observation - SO group
Behavioral: Nature Observation (NO) — The video-clip consisted of a 16 min nature movie in cycles of one-minute observation and pausing 30 s, equivalent to the timing of RMs performed by groups UL and SO
  Arms: (Nature observation -NO group

SUMMARY:
To determine whether there is an ipsilateral transfer of a motor skill from the upper limb to the lower limb

DETAILED DESCRIPTION:
In a single-blind randomized controlled study, 60 healthy subjects randomly participated in one of three single-session interventions: (1) Practicing reaching movement (RM) sequences with the non-dominant left upper limb towards illuminating switches (UL group); (2) Observing the identical sequences of the illuminating switches (Switches Observation (SO) group); and (3) Observing nature movies (Nature Observation (NO) group). Subjects participated in two sessions. The first session included familiarization practice of the motor task, a pretest, a single session intervention (according to group randomization), and a posttest. The second session included a retest, 24 hours after the training.

Recording apparatus used in tests (pretest, posttest, and retest): A custom-made testing device was set up on a rectangular table with a smooth laminated tabletop of 105 cm × 80 cm and adjustable height. Five switch-led units of 5 cm × 8 cm × 5 cm, each composed of a large push-button switch and a red light-emitting diode (LED), attached to the tabletop in a 38-cm radius half circle, successively numbered from 1 to 5. The system was operated by a desktop computer, interfaced with a data acquisition card of LABVIEW software. The algorithm allowed parameters selection of LED activation (illumination) sequence, duration of RM, the delay between RMs, and the number of RM repetitions. Activation of a specific unit LED was a cue for the subject to reach toward that unit and press the push-button switch. Reaching toward the switch of an activated unit deactivated it, and the response time, between the activated and deactivated LED, was recorded.

For testing the leg performance, subjects sat on a custom-designed plinth with a solid back support in front of the apparatus at the same height as the tabletop, hence they could perform the RM sequence with the leg. At the starting position, the heel was placed on the edge of the table in front of switch 3, so when the left heel touched switch 3, the knee reached 30° flexion.

Training conditions: In each of the UL, SO, and NO groups, a 16-minute single-session intervention was conducted. The initial testing position of the subjects during the intervention was sitting on a chair with solid back support, hips, and knees flexed 90°, in front of the apparatus used for the tests. The starting position of the UL group was placing the left fist on the edge of the table in front of the subject's chest (parallel to switch 3) so that they could reach and touch switch 3 with their third left metacarpal. The UL group was instructed to reach with the left UL from the starting position as fast and accurately as possible to the illuminating switch, press it, and return to the starting position, while the fist must remain in contact with the table. They were not notified about the sequence. The subjects performed RMs toward the units that were activated in the same order as the tested sequence 1-4-3-5-4-2, and with an activation duration and delay of 1 s. The practice included 16 blocks, each consisting of 30 RM with a 30 s pause after each block (Fig. 1b). The SO group was instructed to observe the illuminating switches while avoiding moving. The subjects observed RMs toward the units that were activated in the same order as the practiced sequence 1-4-3-5-4-2, also with an activation duration and delay of 1 s and 30 s pause after each block. The NO group was instructed to observe a video clip while avoiding moving. The video clip consisted of a 16 min nature movie in cycles of one-minute observation and pausing 30 s, equivalent to the timing of RMs performed by groups UL and SO.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (self report)
* right hand dominant

Exclusion Criteria:

• musculoskeletal or neurological deficits interfering with task performance (proper upper limb and lower limb reaching performance)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Response Time (msec.) | Pretest - before the training session, posttest - immediately after the training session
  Change in response time (msec.) from pretest to posttest. Activation of a specific unit LED was a cue for the subject to reach toward that unit and press the push-button switch. Reaching toward the switch of an activated unit deactivated it, and the response time, between the activated and deactivated LED, was recorded. Improved motor performance was indicated by a shorter Response Time
Response Time (msec.) | Posttest - immediately after the training session, retest - 24 hours after the training session
  Change in response time (msec.) from posttest to retest. Activation of a specific unit LED was a cue for the subject to reach toward that unit and press the push-button switch. Reaching toward the switch of an activated unit deactivated it, and the response time, between the activated and deactivated LED, was recorded. Improved motor performance was indicated by a shorter Response Time
Response Time (msec.) | Pretest - before the training session, retest - 24 hours after the training session
  Change in response time (msec.) from pretest to retest. Activation of a specific unit LED was a cue for the subject to reach toward that unit and press the push-button switch. Reaching toward the switch of an activated unit deactivated it, and the response time, between the activated and deactivated LED, was recorded. Improved motor performance was indicated by a shorter Response Time

SECONDARY OUTCOMES:
% of fails | Pretest - before the training session, posttest - immediately after the training session
  Change in the % of fails from pretest to posttest. Fails were considered when touching the activated unit-related switch within 1 s. Improved motor performance was indicated by a lower % of fails
% of fails | Posttest - immediately after the training session, retest - 24 hours after the training session
  Change in the % of fails from posttest to retest. Fails were considered when touching the activated unit-related switch within 1 s. Improved motor performance was indicated by a lower % of fails
% of fails | Pretest - before the training session, retest - 24 hours after the training session
  Change in the % of fails from pretest to retest. Fails were considered when touching the activated unit-related switch within 1 s. Improved motor performance was indicated by a lower % of fails

CONTACTS AND LOCATIONS:
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: No
The datasets (Study Protocol, Statistical Analysis Plan, Informed Consent Form, Analytic Code generated during and/or analyzed during the current study) will be available from the corresponding author upon reasonable request.